CLINICAL TRIAL: NCT07343648
Title: Assessment of Antithyroglobulin Antibody Levels Among Diabetic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naira Ali Mohammed Soliman, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: antithyroglobulinAb in DM
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: patients with established diagnosis with diabetes mellitus
- control group: normal individual

SUMMARY:
Assessment of antithyroglobulin antibody (anti Tg) level among diabetic patients explores the intersection between autoimmune thyroid disease and diabetes mellitus. Autoimmune thyroiditis and diabetes frequently coexist, and anti Tg is one of the main markers used to document thyroid autoimmunity.(1,2) Thyroglobulin is a large iodinated glycoprotein produced by thyroid and serves as the precursor for thyroid hormone synthesis. Damage to thyroid tissue in autoimmune thyroiditis leads to production of autoantibodies against thyroglobulin (Tg)(1,3). Anti Tg is therefore considered serologic hallmarks of autoimmune thyroiditis. The presence of this antibody may also be used to monitor thyroid damage progression and predict the development of overt hypothyroidism in at risk populations(1,3).

Type 1 diabetes mellitus (T1DM) is an organ specific autoimmune. Because of shared genetic susceptibility and overlapping immune mechanisms, patients with T1DM have a markedly increased prevalence of autoimmune thyroiditis compared with the general population. International guidelines support routine screening for thyroid autoantibodies and thyroid function in T1DM to enable early detection of subclinical thyroid dysfunction(2,4).

. A study reported that, among 60 T1DM patients without known thyroid disease, 16.7% were positive for anti Tg, and subclinical or overt hypothyroidism was present in a substantial fraction of this antibody positive individuals. Other series similarly show that thyroid autoantibodies are common in T1DM and that their presence predicts later thyroid dysfunction. (5,6).

Increasing evidence indicates that type 2 diabetes mellitus (T2DM) is also associated with a higher prevalence of thyroid autoantibodies than nondiabetic controls in many studies(1,7). In a study including 72 T2DM patients, 20.8% had either anti TPO or anti Tg positivity, and 8.3% had isolated anti Tg antibodies, with rates comparable to or higher than those reported in regional control populations. A study of female T2DM patients found anti Tg in 61.3% of cases compared with no positives in the control group, and more than half of hypothyroid diabetic patients had anti Tg positivity, suggesting a significant autoimmune contribution to thyroid dysfunction in some T2DM cohorts. (2,8).

Autoimmune clustering means that diabetic patients, are predisposed to additional organ specific autoimmune diseases, including autoimmune thyroiditis. Screening for anti Tg provides a more complete picture of thyroid autoimmunity. (2,8)

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-80 years, both genders.
* established diagnosis with diabetes mellitus

Exclusion Criteria:

* History of thyroid disease
* Prior thyroid surgery
* Current thyroid replacement or anti-thyroid medication
* Use (within last 3 months) of drugs known to affect thyroid function or antibodies
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with established diagnosis with diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
the levels of anti-thyroglobulin (anti-Tg) antibodies among diabetic patients . | baseline
  the levels of anti-thyroglobulin (anti-Tg) antibodies among diabetic patients .